CLINICAL TRIAL: NCT00113425
Title: Photodynamic Therapy in the Treatment of Acne Vulgaris
Brief Title: Non-cutting Laser Therapy in the Treatment of Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey S. Orringer, Professor of Dermatology, University of Michigan, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 548
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Acne Vulgaris
Keywords: non-ablative laser; acne; photosensitizer; photodynamic therapy
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Therapy (Experimental): V-Beam laser, Candela Corp., 595 nm wavelength
  Interventions: Device: V-Beam laser, Candela Corp., 595 nm wavelength
- Control (No Intervention): Untreated

INTERVENTIONS:
Device: V-Beam laser, Candela Corp., 595 nm wavelength — Subjects will receive a series of up to 6 laser therapy sessions with a treatment interval of from approximately 1 to 4 weeks. In all cases, laser treatment parameters will be within the guidelines normally used clinically with the V-Beam laser, and thus fluences used will not exceed 15 J/cm2.
  Arms: Laser Therapy

SUMMARY:
The purpose of this research project is to study the effect of non-ablative (non-cutting) laser therapy, a technique that uses laser energy to try to improve the appearance of the skin. This type of laser treatment creates changes in a layer of the skin called the dermis without causing an open wound in the skin. The use of non-ablative laser therapy, together with application of a photo-sensitizer (substance that makes the skin more sensitive to light), may improve the appearance of acne. The idea behind the photo-sensitizer is that it is supposed to make the laser more effective than using just the laser alone. It is not yet clear how much improvement can be seen with these treatments or exactly how the skin's response causes these improvements. In this study, we are interested in learning how well such a laser works to improve the symptoms of acne, as well as how much the photo-sensitizer actually enhances the efficacy of the laser.

DETAILED DESCRIPTION:
Acne vulgaris remains among the most common cutaneous disorders, impacting the vast majority of people at some point during their lives. It is associated with significant psychosocial morbidity, and there remains the need for efficacious and low risk therapeutic options.

Recently, the FDA has approved various lasers for the treatment of acne. However, few randomized, controlled clinical trials have been performed. In addition, the use of topical photosensitizers preceding laser therapy for acne has also been examined in a preliminary way with some initial evidence of efficacy. However, these small trials have primarily focused on back acne and have included modest numbers of subjects. Photodynamic therapy for facial acne is being performed by physicians across the country but little objective data regarding this practice is available.

We propose to evaluate the efficacy and confirm the safety of pulsed dye laser therapy (V-Beam laser, Candela Corp., Wayland, MA, 595 nm wavelength) used in conjunction with a topical photosensitizer in the treatment of acne vulgaris. This is a split-face comparison study in which one half of the face will be treated with photo-sensitizer and laser, and the contralateral side will be left untreated. Because one proposed mechanism of action for such treatments includes altered sebaceous gland activity, we also seek to examine the effects of this treatment on cutaneous sebum production.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years or older of either gender and of any racial/ethnic group.
* Presence of clinically-evident facial acne.
* Subjects must be in generally good health.
* Subjects must be able and willing to comply with the requirements of the protocol.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Oral retinoid (Accutane) use within 6 months of entry into the study.
* Systemic acne therapies (oral antibiotics) within 4 weeks of entry into the study.
* Topical acne therapies (retinoids, antibiotics) within 2 weeks of entry into the study.
* Microdermabrasion or superficial chemical peels at the sites to be treated within 2 months of entry into the study.
* Subjects with a history of dermabrasion or laser resurfacing at the sites to be treated.
* Use of topical lipid absorbing substances (Clinac AC) within 2 weeks of entry into the study.
* Non-compliant subjects.
* Subjects with a significant medical history or concurrent illness/condition which the investigator(s) feel is not safe for study participation.
* Subjects using alcohol-based topical solutions or "exfoliating" agents within 2 weeks of entry into the study.
* Subjects with a history of very frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
* History of keloid (excessive scar) formation for subjects undergoing biopsies.
* Pregnant or nursing females.
* Subjects with known allergy or hypersensitivity to topical photosensitizing agents.
* Subjects with known photosensitivity disorders felt by the investigators to preclude safe inclusion in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Patients were randomized to receive topical photosensitizer applications followed by pulsed dye laser therapy to one side of the face while the contralateral side of the face remained untreated, thus serving as an internal control.
Period: Overall Study
Arm/Group | All Study Participants
Started | 44
Completed | 29
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Treated Group Pulsed Dye Laser Therapy and Untreated Group: Patients were randomized to receive topical photosensitizer applications followed by pulsed dye laser therapy to one side of the face and the contralateral side of the face remained untreated, thus serving as an internal control.
Arm/Group | Treated Group Pulsed Dye Laser Therapy and Untreated Group
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.41 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5
  Black / African American | 3
  Caucasian | 30
  Hispanic, Latina | 2
  Middle Eastern | 2
  More than one race | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Papule Acne Lesions at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: papule acne lesions
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
papule acne lesions
  Change from Baseline on Treated Side | -4.63 [-7.43 to -1.83]
  Change from Baseline on Untreated Side | -0.13 [-2.83 to 2.57]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in papule acne lesions for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.01, paired t-test, 2-sided

2. Primary Outcome: Change From Baseline in Pustule Acne Lesions at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: pustule acne lesions
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
pustule acne lesions
  Change from Baseline on Treated Side | -1.80 [-5.05 to 1.45]
  Change from Baseline on Untreated Side | -1.20 [-4.49 to 2.09]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in pustule acne lesions for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.43, paired t-test, 2-sided

3. Primary Outcome: Change From Baseline in Cysts at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: cysts
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
cysts
  Change from Baseline on Treated Side | 0.10 [-0.35 to 0.55]
  Change from Baseline on Untreated Side | 0.07 [-0.30 to 0.43]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in cysts for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.79, paired t-test, 2-sided

4. Primary Outcome: Change From Baseline in Closed Comedones at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: closed comedones
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
closed comedones
  Change from Baseline on Treated Side | -5.07 [-10.53 to 0.40]
  Change from Baseline on Untreated Side | -1.17 [-7.52 to 5.19]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in closed comedones for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.10, paired t-test, 2-sided

5. Primary Outcome: Change From Baseline in Open Comedones at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: open comedones
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
open comedones
  Change from Baseline on Treated Side | -1.00 [-6.37 to 4.37]
  Change from Baseline on Untreated Side | -0.63 [-6.01 to 4.75]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in open comedones for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.73, paired t-test, 2-sided

6. Primary Outcome: Change From Baseline in Erythematous Macules at Week 10
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: erythematous macules
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
erythematous macules
  Change from Baseline on Treated Side | -1.88 [-7.73 to 3.97]
  Change from Baseline on Untreated Side | 1.28 [-4.66 to 7.22]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in erythematous macules for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.02, paired t-test, 2-sided

7. Primary Outcome: Change From Baseline in Acne Severity at Week 10
Description: The Leeds scale is a 12-point ordinal photonumeric global acne severity scale where a rating of 1 denotes the mildest acne and a rating of 12 represents the most severe.
Time Frame: Baseline and Week 10
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
units on a scale
  Change from Baseline on Treated Side | -0.90 [-1.30 to -0.50]
  Change from Baseline on Untreated Side | -0.30 [-0.65 to 0.05]
Statistical Analysis 1: Comparison: All Study Participants; Null Hypothesis = There is no difference between change from baseline in acne severity for the treated side of the face compared to the change from baseline for the untreated side of the face in all patients; Test type: Superiority or Other; p = 0.003, paired t-test, 2-sided

8. Secondary Outcome: Change From Baseline in Papule Acne Lesions at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: papule acne lesions
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
papule acne lesions
  Change from Baseline on Treated Side | -1.79 [-5.98 to 2.39]
  Change from Baseline on Untreated Side | -0.97 [-4.32 to 2.39]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.62, paired t-test, 2-sided

9. Secondary Outcome: Change From Baseline in Pustule Acne Lesions at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: pustule acne lesions
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
pustule acne lesions
  Change from Baseline on Treated Side | -2.72 [-6.65 to 1.20]
  Change from Baseline on Untreated Side | -2.62 [-6.25 to 1.01]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.85, paired t-test, 2-sided

10. Secondary Outcome: Change From Baseline in Cysts at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: cysts
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
cysts
  Change from Baseline on Treated Side | 0.38 [-0.20 to 0.96]
  Change from Baseline on Untreated Side | 0.24 [-0.33 to 0.82]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.49, paired t-test, 2-sided

11. Secondary Outcome: Change From Baseline in Closed Comedones at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: closed comedones
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
closed comedones
  Change from Baseline on Treated Side | -6.97 [-13.30 to -0.63]
  Change from Baseline on Untreated Side | -4.07 [-9.12 to 0.98]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.21, paired t-test, 2-sided

12. Secondary Outcome: Change From Baseline in Open Comedones at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: open comedones
Arm/Group | All Study Participants
Number analyzed (Participants) | 29
open comedones
  Change from Baseline on Treated Side | -4.79 [-11.62 to 2.04]
  Change from Baseline on Untreated Side | -6.79 [-13.88 to 0.29]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.27, paired t-test, 2-sided

13. Secondary Outcome: Change From Baseline in Erythematous Macules at Week 16
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: erythematous macules
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
erythematous macules
  Change from Baseline on Treated Side | -5.89 [-12.12 to 0.34]
  Change from Baseline on Untreated Side | -2.50 [-8.85 to 3.85]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.04, paired t-test, 2-sided

14. Secondary Outcome: Change From Baseline in Acne Severity at Week 16
Description: as for outcome 7
Time Frame: Baseline and Week 16
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
units on a scale
  Change from Baseline on Treated Side | -1.07 [-1.69 to -0.45]
  Change from Baseline on Untreated Side | -0.52 [-1.07 to 0.04]
Statistical Analysis 1: Comparison: All Study Participants; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.01, paired t-test, 2-sided

ADVERSE EVENTS:
Groups:
- Treated Group Pulsed Dye Laser Therapy: Patients were randomized to receive topical photosensitizer applications followed by pulsed dye laser therapy to one side of the face.
- Untreated Group Control: The contralateral side of the face remained untreated, thus serving as an internal control.
Arm/Group | Treated Group Pulsed Dye Laser Therapy | Untreated Group Control
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 5/44 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Group Pulsed Dye Laser Therapy (N=44) | Untreated Group Control (N=44)
Mild Peeling (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Transient Postinflammatory Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes